CLINICAL TRIAL: NCT03904160
Title: Web-based Personal or Peer Group Weight Management Study
Acronym: PERGROUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Päivi Korhonen, Professor of General Practice, University of Turku
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 10618012017
Record Dates: First submitted 2018-10-20; First posted 2019-04-05 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Overweight and Obesity; Cardiovascular Risk Factors; Quality of Life; Work Ability
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nurse-lead group (Sham Comparator): Nurse-lead sessions for weight management. Ten sessions lasting 90 minutes each in three groups of 10-14 participants. Each session comprise education about healthy diet, psychoeducation and discussions.
  Interventions: Behavioral: Weight management
- Web-based group (Experimental): Web-based weight management system with peer-based conversation possibility. Three groups of 10-14 participants who gather together for three nurse-lead sessions in the weeks 0, 5, and 12. The web-based program can be used for a year.
  Interventions: Behavioral: Weight management
- Web-based personal (Experimental): Web-based weight management system with conversation possibility with the nurse for 12 weeks. Altogether 37 participants who can use the web-based weight management system for one year.
  Interventions: Behavioral: Weight management

INTERVENTIONS:
Behavioral: Weight management — Please see the arm descriptions.

SUMMARY:
The PERGROUP trial aims to investigate whether Web-based personal or Web-based group counselling weight management program can help to achieve lifestyle changes needed for weight loss and improvement in quality of life and cardiovascular risk factors. The control group is the traditional nurse-lead weight management group counselling.

DETAILED DESCRIPTION:
In this study, efficacy of two web-based weight management systems will be compared to a traditional nurse-lead sessions for weight management.

Ten nurse-lead group counselling sessions lasting 90 minutes each will be conducted in three groups of 10-14 participants. Each session comprise education about healthy diet, psychoeducation and discussions.

The web-based group counselling program offers informative weight management system with peer-based conversation possibility. Three groups of 10-14 participants who gather together for three nurse-lead sessions in the weeks 0, 5, and 12. The web-based program can be used for a year.

The web-based personal counselling program offers informative weight management system with conversation possibility with the nurse for 12 weeks. Altogether 37 participants are enrolled and they can use the web-based weight management system for one year.

In each intervention arm, intervention and counselling provided by the study nurses last for three months. Among all participants, weight loss, cardiometabolic data, information of lifestyle and quality of life will be measured at baseline, after the nurse-lead intervention (three months) and 12 months from the baseline.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 25 kg/m2 or higher

Exclusion Criteria:

* pregnancy
* active cancer
* acute cardiovascular event less than three months before
* untreated thyroid disease
* systematic corticosteroid medication
* anorexia or bulimia
* impaired communication ability

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 109 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
The number of participants who obtained and maintained a weight loss of at least 5% at 12 months | From baseline to 12 months
  The number of participants who obtained and maintained a weight loss of at least 5% at 12 months

SECONDARY OUTCOMES:
Work ability | From baseline to 12 months
  The percentage of participants in whom weight management intervention will be associated with participants´ Work Ability Score (WAS). The total score range is 0 to 10 with higher value representing better work ability.
Overall quality of life measured by the Eurohis instrument | From baseline to 12 months
  The number of participants in whom weight management intervention will be associated with quality of life assessed by the Eurohis instrument. Mean change from baseline in frequencies of reported problems will be reported.
Health-related quality of life measured with the EuroQol instrument. | From baseline to 12 months
  The number of participants in whom weight management intervention will be associated with quality of life assessed by the EuroQol instrument. Mean change from baseline in frequencies of reported problems will be reported.
Change in systolic blood pressure in mmHg | From baseline to 12 months
  Change in systolic blood pressure in mmHg
Change in diastolic blood pressure in mmHg | From baseline to 12 months
  Change in diastolic blood pressure in mmHg
Change in waist circumference in centimeters | From baseline to 12 months
  Change in waist circumference in centimeters
Change in weight in kilograms | From baseline to 12 months
  Change in weight in kilograms
Change in body mass index. | From baseline to 12 months
  Change in body mass index. Weight and height will be combined to report body mass index in kg/m2
Change in body fat percentage | From baseline to 12 months
  Change in body fat percentage
Change in plasma total cholesterol in mmol/l | From baseline to 12 months
  Change in plasma total cholesterol in mmol/l
Change in plasma high-density lipoprotein cholesterol in mmol/l | From baseline to 12 months
  Change in plasma high-density lipoprotein cholesterol in mmol/l
Change in plasma low-density lipoprotein cholesterol in mmol/l | From baseline to 12 months
  Change in plasma low-density lipoprotein cholesterol in mmol/l
Change in plasma triglycerides in mmol/l | From baseline to 12 months
  Change in plasma triglycerides in mmol/l
Change in plasma fasting glucose in mmol/l | From baseline to 12 months
  Change in plasma fasting glucose in mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Lehtimäki, Study Chair — Satakunta Heart District
Locations (1):
- Satakunta Heart District, Pori, Finland

IPD SHARING:
Plan to Share IPD: Undecided